CLINICAL TRIAL: NCT03186872
Title: Improving Quality of Care With a Digital Behavioral Program in IBD Patient Centered Medical Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Mount Sinai Hospital, New York (Other)
Responsible Party: Principal Investigator, Marc Schwartz, Assistant Professor of Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PRO17020464
Record Dates: First submitted 2017-06-06; First posted 2017-06-14 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Anxiety; Irritable Bowel Disease
MeSH Terms: conditions — Anxiety Disorders; Irritable Bowel Syndrome | interventions — nano-lantern protein

STUDY DESIGN:
Intervention Model Description: Comparison between cognitive behavioral app and care as usual.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Care as usual (No Intervention): Participants randomized to this group will continue to see the IBD medical home team as usual
- Digital behavioral program app (Experimental): Participants randomized to this group will see the IBD medical home team and will utilize the cognitive behavioral app as the intervention.
  Interventions: Behavioral: Digital behavioral program app

INTERVENTIONS:
Behavioral: Digital behavioral program app — mobile app utilizing cognitive behavioral techniques to help alleviate anxiety
  Other Names: Lantern
  Arms: Digital behavioral program app

SUMMARY:
Anxiety disorders and depression are more prevalent in patients living with inflammatory bowel disease (IBD) than in healthy controls. Approximately 40% of IBD patients have elevated anxiety. Given the robust effectiveness of cognitive behavioral approaches for anxiety disorders and the paucity or mixed findings of cognitive behavioral approaches for anxiety in IBD, an integrated behavioral approach and combining face to face and online cognitive behavioral modalities is recommended for IBD patients with anxiety.

DETAILED DESCRIPTION:
If the patient is eligible for, interested in, and consents to, participating in this study, the social worker will use the randomization program (social worker remains blind to random assignment until the moment this group assignment is delivered to the patient) to determine to which group the patient is randomized. The Social Worker will provide the patient's MRN, name, date of birth and contact information to the UPMC research team. The UPMC research team will generate a unique ID for each patient. Lantern is a behavioral health app that is used to help people manage their stress and anxiety. There are many modules that the subjects will be offered through the course of Lantern. There is a coach available to the subject who will guide the subject through the modules and be available for check-ins.For those patients that are randomized to Lantern at baseline, they will be provided a postcard with a sign up code so they can sign up directly on their mobile device. The PCMH research assistant will assign a study ID at the time of consent and study enrollment and enter this into the UPMC study database. Once patient is in Lantern, they are assigned a Lantern User ID. The Lantern User ID along with DOB and name will be sent to the UPMC research team through a secure VPN connection so that a crosswalk can be created in the UPMC study database that links their study IDs and Lantern User IDs. Patients will be recommended to start and use the anxiety management program to help address their anxiety/stress symptoms. The techniques to try are available for participants to access at any time. The coaches are not therapists, but are there to provide information and encouragement to the patient. To keep confidentiality, the coach only knows the first name of the patient. The coordinator of the coaches has access to the patient's identifying information if the patient has an escalation in distress/anxiety that needs to be addressed. This information will be passed to the PI when necessary as part of the escalation procedures (as outlined above in Section 2.5.2 and in the attachments- Escalation Procedure). The personally identifying information is held internally within the Amazon web services at Lantern. The coaches for the patients have access to an internal Coaching Portal where they have a dashboard for each of their users. This dashboard includes all information that the user inputs into the Lantern program, including both their direct messages to coaches and all content they complete in the program. Coaches receive a notification when users complete a path in the program or send them a message, which prompts their response to the individual (See Other Attachments - Example Messages from Lantern Coaches to read examples of how the coach interacts with the user as well as Sample Lantern Content.) The 6 core components include:1. Education and awareness about stress and how thoughts, emotions, and behaviors are interrelated. This provides the rationale of the cognitive behavioral model. In this unit, patients will learn how you can change your thoughts and behaviors to change your emotions. 2. Relaxation - patients learn several empirically supported relaxation techniques to manage stress/anxiety. 3. Thoughts - This unit is about the stories we tell ourselves and how these stories determine our mood and help us decide what actions we will take. This component also guides patients how to challenge their assumptions about these thoughts/stories to create new stories.4. Behavior Change and Exposure - patients will learn how to avoid things that contribute to stress and identify adaptive coping activities. Through learning the principle of exposure, patients learn how exposing themselves to anxiety provoking situations can help to overcome anxiety in the long-term.5. Mindfulness - This unit is about taking a step back from our thoughts and feelings to interrupt the thoughts-feelings-behaviors cycle. Several mindfulness exercises are offered so the patient can find the type that feels best for them.6. Habit formation/Maintaining skills - patients will reflect on what they have learned and work on making a habit out of the most effective techniques.Lantern, the third-party program provider, will collect de-identified usage data (e.g., progression through the program, frequency of messages to coaches, and techniques completed) and quantitative data (e.g., anxiety score responses) as the patients' progress through the program. Lantern internally has a database that tracks user progress through the programs, so they understand how patients have moved through the program. This de-identified data will be sent to the UPMC study staff coded only with the patient's unique ID. At several time points, Lantern will push self-report validated questionnaires (e.g., GAD7) to patients enrolled in Lantern via their Qualtrics account. Lantern's Qualtrics Account is a third party, HIPAA compliant survey tool. Thrive Network, Inc. has a Business Associate Agreement (BAA) with Lantern's Qualtrics Account and owns all data collected through surveys. Lantern will share this de-identified self-report questionnaire data with the UPMC clinical team using unique Lantern User IDs. Lantern's coaches will not have access to any of the questionnaire data collected via Qualtrics. For those patients randomized to PCMH Behavioral Health control condition at baseline to 3 months, they will receive PCMH care as usual without any skills-based behavior therapy. Standard behavioral health clinical monitoring will continue to occur according to best practice guidelines. Specifically, this means that for patients with a baseline GAD7 > 10 will receive a phone call from a PCMH behavioral health provider to do a mood check at one month after baseline assessment. Regardless of baseline GAD7 score, if the baseline PHQ2 > = 3, a behavioral health provider will conduct the phone call for a mood check at one month follow up. From the baseline PHQ8 assessments, we will extrapolate the PHQ2 to use for clinical decision making to rely on affective components of depression rather than somatic component as this overlaps substantially with inflammatory-related medical conditions. At 3 month study follow-up, patients in both groups will be re-assessed with the study assessment battery (outlined in measures section and in Table x). Non-responders will be re-randomized to an adaptive care strategy. The 3 month GAD7 assessment will be used to determine 'responder' vs. 'non-responder' status. In the Lantern group, patients are defined as 'non-responders' if their 3 month GAD7 is > = 11 or if there is < 4 point reduction on GAD7. These cutoff scores and magnitude of change are based on the literature establishing thresholds for 'treatment response'. We conservatively estimate a 40% non-response rate in Mobile anxiety self-management program group based on CBT for anxiety meta-analyses. In the PCMH Behavioral Health control condition, 'non-responders' are defined as 3 month GAD7 scores increasing by >=3 points from baseline. It's estimated that 1/2 of patients in PCMH (behavioral health WL control) will either be responders or remain stable/unchanged based on findings of natural course of in GAD. At 3 months, the Lantern non-responders will be re-randomized to either 1) PCMH care as usual (i.e., this includes individual skills-based behavioral therapy provided by behavioral health providers) or 2) PCMH care as usual + Lantern. The PCMH Behavioral Health Control group non-responders will be re-randomized to either 1) PCMH care as usual or 2) Lantern only. For PCMH care as usual groups, individual CBT will be provided as follows: if 3 month GAD7 > = 15 and/or PHQ2 >=4, the patient will be offered every other week CBT sessions. If 3 month GAD7 and PHQ2 are below these thresholds, then patients will be offered monthly individual CBT sessions. The 'Responders' will continue in their original randomly assigned group (either Lantern or PCMH Behavioral Health control group). All study participants will engage in their respective care approaches for another three-month period and then the same study assessment battery will be re-administered at 6 months. For those patients who were defined as 'responders/stable' at 3 months within the PCMH Behavioral Health Control group, standard behavioral health clinical monitoring will continue. Specifically, if 3 month GAD7 > = 15 and/or 3 month PHQ2 >=3, then a behavioral health provider will call the patient monthly to conduct mood check ins. A subset of participants (12 completers and 12 non-completers)who were offered the stress management app will be asked to participate in an in-depth qualitative phone interview 6 months after enrollment. Participants will be randomly selected and will include those who completed and those who did not complete the program. The interviews will be conducted by research staff contacting the randomly selected subjects. The qualitative interview will explore patient's experience with the program and areas of suggested improvement. All interviews will be audio-recorded and transcribed verbatim. All study participants, regardless of the condition to which they are assigned, will complete the study assessment battery at 9 and 12 months as well.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are seeking medical care at UPMC IBD Patient Centered Medical Home (PCMH); age 21-55; GAD7 score >/= 8, English speaking and capable of understanding the informed consent and providing consent; access to a Smartphone

Exclusion Criteria:

* No psychotherapy within PCMH within past 6 months including with the psychologist• Stable on psychiatric meds for 4 weeks• Personality pathology or PTSD (captured from DSM-V cross cutting symptoms inventory already being used as part of routine care screening in this clinic)• Severe mood disorder (PHQ8 > 14) or evidence of active suicidality or psychosis (brief screen conducted by SWer in clinic using DSM-V cross cutting symptom inventory) to assess for psychosis, etc. will serve as our study screener • No smartphone

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2019-05-29 (Actual); Study Completion 2019-05-29 (Actual)

PRIMARY OUTCOMES:
GAD7 Score (Anxiety) | 12 months
  GAD7 anxiety questionnaires are completed at time points throughout the study.

SECONDARY OUTCOMES:
PHQ-8 (Depression) | 12 months
  The PHQ-8 questionnaire about depression is completed at different time points throughout the study.

OTHER OUTCOMES:
ACE Measure | 12 months
  ACe questionnaire about health and health care is completed at time points throughout the study.
Ulcerative Colitis Activity Index (UCAI)/Harvey Bradshaw (HB) | 12 months
  The UCAI/HB questionnaires about IBD related chronic pain are completed at time points throughout the study. The subject completes the appropriate questionnaire based on IBD diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Schwartz, MD, Principal Investigator — University of Pittsburgh Medical Center; Eva Szigethy, MD, PhD, Study Director — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
IPD data will not be shared. Data is shared at the aggregate level.

REFERENCES:
- [Derived] Oser M, Wallace ML, Solano F, Szigethy EM. Guided Digital Cognitive Behavioral Program for Anxiety in Primary Care: Propensity-Matched Controlled Trial. JMIR Ment Health. 2019 Apr 4;6(4):e11981. doi: 10.2196/11981. PMID 30946022